CLINICAL TRIAL: NCT03922516
Title: Accuracy of Ultra-Low-Dose-CT (ULDCT) of the Chest Compared to Plain Film in an Unfiltered Emergency Department Patient Cohort
Brief Title: Accuracy of Ultra-Low-Dose-CT of the Chest Compared to Plain Film in an Unfiltered Emergency Department Patient Cohort
Acronym: UP-Chest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Siemens AG (Industry)
Responsible Party: Principal Investigator, Prof Helmut Ringl, MD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: EK-Nr. 2254/2018
Record Dates: First submitted 2019-04-17; First posted 2019-04-22 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Chest Pain; Cough; Thoracic Diseases; Lung Diseases
MeSH Terms: conditions — Chest Pain; Cough; Thoracic Diseases; Lung Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reporting order: Plain Film - ULDCT (Other): The plain film of half the participants (randomized) will be submitted for reporting by a radiologist as a first imaging method. After finishing this report, the same radiologist will assess the ULDCT of this participant. In this second report, the findings of both examinations will be summarized, and a second report will be filed.
  Emergency physicians will first receive the report for the plain film of the chest and will be asked for the diagnosis and its probability. Next, the report for ULDCT will be presented to them. Again, diagnosis and probabilities will be documented.
  Interventions: Diagnostic Test: ULDCT
- Reporting order: ULDCT - Plain Film (Other): For half the participants (randomized) radiologists will first receive the data from ULDCT of the chest and write a report. Subsequently, they will receive the data from the plain film of the chest and may expand their report (explicitly separated).
  Emergency physicians will first receive the report for the ULDCT of the chest and will be asked for probabilities of the nine most frequent diagnoses in chest-imaging plus "other". Next, they will be presented with the report for the plain film and will again be asked to give an estimation of the probabilities for the same diagnoses as before.
  Interventions: Diagnostic Test: ULDCT

INTERVENTIONS:
Diagnostic Test: ULDCT — Ultra-Low-Dose-CT (ULDCT) of the chest using tin filters with third-generation dual-energy CT devices. The projected dose used will be approximately 0.2 mSv per ULDCT of the chest.

SUMMARY:
This trial compares the accuracy provided by plain film as well as ultra-low-dose-computed-tomography (ULDCT) of the chest. It also aims to analyze differences in diagnostic confidence and therapeutic consequence offered by these two imaging modalities.

DETAILED DESCRIPTION:
For nearly a century, chest X-ray (plain film, projectional radiography) has been the established primary imaging modality for patients with acute chest pain, suspected pneumonia, and / or acute dyspnoea in the diagnostic pathway of emergency departments, although the sensitivity and specificity of this X-ray technique are moderate.

The widespread availability and use of chest X-ray is due to the low acquisition and operating costs for projectional radiography equipment, the short examination time, and the very low radiation exposure. In addition, projectional radiography of the chest often serves as a guide for further, more sensitive, diagnostical procedures. However, these advantages are partially offset by the disadvantages inherent to projectional methods: anatomical structures may superpose or mask pathological structures. As a result, some areas of the lung may be obscured, and assessment may therefore be limited.

Whereas computed tomography was reserved for certain clinical questions over the last few decades, and, in most cases, served as a second imaging approach after plain film radiography, it has increasingly evolved as a primary imaging modality for several indications (e.g., suspicion of pulmonary embolism, highly suspected aortic dissection). This rise of computed tomography was due not only to its significant advantage of no superposition, but also partly driven by the marked reduction in radiation dose needed without sacrificing image quality. This was driven by the development of new detectors, modulation of tube current and voltage, as well as iterative reconstruction techniques. As a result, recent computed tomography scanners currently offer not only a more precise visualization of differences in tissue-attenuation and the significant advantage of the absence of artefacts due to superposition, but also allow for imaging with a considerably reduced radiation dosage compared to older scanners. Therefore, computed tomography may now be utilized as screening method in specific indications that carry an increased risk of certain pathologies (e.g., in long-time smokers). The introduction of the latest generation of computed tomography devices about three years ago allowed for an even further reduction in dose by filtering out low-energy photons using a tin filter, which offers the possibility of a reduction in radiation dose by another 50 % or more for established CT indications. For specific indications (e.g., lung nodules in follow-up), the radiation dose may even be reduced to a tenth or one-hundredth of a standard-dose CT (SDCT).

The current reference dose-length-product (DLP) in Germany for thoracic standard-dose CT (SDCT) is ~350 mGycm (effective dose ~6 mSv) and, for thoracic low-dose-CT (LDCT / HR-CT), ~100 mGycm (effective dose ~1.7 mSv). However, the latest devices (third-generation dual-energy CT) provide the opportunity to considerably reduce the reference dose of thoracic low-dose CT. In the current literature, these scans are referred to as Ultra-Low-Dose-CT (ULDCT) and are usually associated with a radiation dosage of 0.14 to 0.5 mSv. For this dose range, no standardized reference values have been published as yet.

The limiting factors of ULDCT are quantum noise, loss of spatial resolution, and other image artefacts. Therefore, careful selection of appropriate CT protocols and dosage is mandatory in order to achieve sufficient image quality to answer the respective diagnostic question.

Several papers have been published on the subject of ULDCT, which are dedicated to the comparison of ULDCT with LDCT and/or SDCT. These papers conclude that this technology may be used with sufficient sensitivity and specificity for indications such as dyspnea, emphysema, or lung nodules. Due to the potential to reduce the radiation dose to less than 1/30 of a standard-dose CT while still providing acceptable image quality with the latest generation of devices, ULDCT of the chest is emerging as an interesting alternative to conventional chest X-ray.

To the best of the authors' knowledge, there are currently no studies comparing and evaluating ultra-low-dose-CT as a primary imaging alternative to chest X-ray in emergency department patients.

This study aims to compare ULDCT and plain film of the chest with regard to their accuracy in an unfiltered patient cohort of an emergency department. For this purpose, the investigator's ULDCT protocol will use the lowest possible dose at which image quality is diagnostically sufficient (approximately 0.2 mSv effective dose). This corresponds to less than 1/30 of the radiation dose of a standard-dose CT of the chest and to only about 2.5 times the dose of a chest X-ray in two views. This dose is equal to less than a month of natural background radiation in Austria and less than the radiation exposure on an intercontinental flight.

In addition to the accuracy of ULDCT of the chest compared to plain film of the chest, this trial also aims to analyze the clinical relevance of both methods by assessing the respective impact on final diagnosis, as well as possible changes in therapy.

ELIGIBILITY:
Inclusion Criteria:

* all patients who are assigned to a clinically indicated chest X-ray by the emergency department of Vienna General Hospital
* ability to provide informed consent
* informed consent after detailed patient briefing

Exclusion Criteria:

* the emergency departments assessment of a critical clinical condition oppose an examination with both modalities (ULDCT of the chest, chest X-ray)
* assigned to chest X-ray as follow-up
* women with positive ß-HCG-test

Ages: 18 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of ultra-low-dose-CT of the chest and plain film of the chest | 1 year
  Initial radiologic diagnostic accuracy of both methods will be assessed by analyzing the number of reports that are changed after the images of the second modality become available to the radiologist in Arm 1 compared to Arm 2.
  In a final approach, the diagnostic accuracy will be analyzed by retrospectively comparing all reports with the gold standard, which will be built from all available patient data at the end of the study, including all follow-up imaging studies and laboratory tests.

SECONDARY OUTCOMES:
Sensitivity and Specificity of ULDCT and plain film | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of change in radiological diagnosis | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of change in emergency physician's diagnosis | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of change in (planned) therapeutic course of action by emergency physician | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of accidental diagnosis in ULDCT and plain film | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of additional diagnostic imaging needed | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Frequency of unclear reports in ULDCT and plain film | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Diagnostic confidence in ULDCT and plain film by radiologist | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"
Diagnostic confidence in ULDCT and plain film by emergency physician | 1 year
  Comparison between the two arms "ULDCT - Plain Film" and "Plain Film - ULDCT"

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Ringl, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Vienna General Hospital - Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van der Aalst CM, Ten Haaf K, de Koning HJ. Lung cancer screening: latest developments and unanswered questions. Lancet Respir Med. 2016 Sep;4(9):749-761. doi: 10.1016/S2213-2600(16)30200-4. PMID 27599248
- [Background] Andronikou S, Lambert E, Halton J, Hilder L, Crumley I, Lyttle MD, Kosack C. Guidelines for the use of chest radiographs in community-acquired pneumonia in children and adolescents. Pediatr Radiol. 2017 Oct;47(11):1405-1411. doi: 10.1007/s00247-017-3944-4. Epub 2017 Sep 21. PMID 29043422
- [Background] Radiation Emissions from Computed Tomography: A Review of the Risk of Cancer and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2014 Jun 4. Available from http://www.ncbi.nlm.nih.gov/books/NBK263458/ PMID 25535640
- [Background] Berrington de Gonzalez A, Mahesh M, Kim KP, Bhargavan M, Lewis R, Mettler F, Land C. Projected cancer risks from computed tomographic scans performed in the United States in 2007. Arch Intern Med. 2009 Dec 14;169(22):2071-7. doi: 10.1001/archinternmed.2009.440. PMID 20008689
- [Background] Braun FM, Johnson TR, Sommer WH, Thierfelder KM, Meinel FG. Chest CT using spectral filtration: radiation dose, image quality, and spectrum of clinical utility. Eur Radiol. 2015 Jun;25(6):1598-606. doi: 10.1007/s00330-014-3559-1. Epub 2014 Dec 17. PMID 25515204
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] Cardinale L, Priola AM, Moretti F, Volpicelli G. Effectiveness of chest radiography, lung ultrasound and thoracic computed tomography in the diagnosis of congestive heart failure. World J Radiol. 2014 Jun 28;6(6):230-7. doi: 10.4329/wjr.v6.i6.230. PMID 24976926
- [Background] Chalmers JD. The Modern Diagnostic Approach to Community-Acquired Pneumonia in Adults. Semin Respir Crit Care Med. 2016 Dec;37(6):876-885. doi: 10.1055/s-0036-1592125. Epub 2016 Dec 13. PMID 27960211
- [Background] Chawla A, Rajendran S, Yung WH, Babu SB, Peh WC. Chest radiography in acute aortic syndrome: pearls and pitfalls. Emerg Radiol. 2016 Aug;23(4):405-12. doi: 10.1007/s10140-016-1415-0. Epub 2016 Jun 9. PMID 27282377
- [Background] Fintelmann FJ, Gottumukkala RV, McDermott S, Gilman MD, Lennes IT, Shepard JO. Lung Cancer Screening: Why, When, and How? Radiol Clin North Am. 2017 Nov;55(6):1163-1181. doi: 10.1016/j.rcl.2017.06.003. PMID 28991558
- [Background] Haubenreisser H, Meyer M, Sudarski S, Allmendinger T, Schoenberg SO, Henzler T. Unenhanced third-generation dual-source chest CT using a tin filter for spectral shaping at 100kVp. Eur J Radiol. 2015 Aug;84(8):1608-1613. doi: 10.1016/j.ejrad.2015.04.018. Epub 2015 Apr 28. PMID 26001437
- [Background] Horeweg N, Scholten ET, de Jong PA, van der Aalst CM, Weenink C, Lammers JW, Nackaerts K, Vliegenthart R, ten Haaf K, Yousaf-Khan UA, Heuvelmans MA, Thunnissen E, Oudkerk M, Mali W, de Koning HJ. Detection of lung cancer through low-dose CT screening (NELSON): a prespecified analysis of screening test performance and interval cancers. Lancet Oncol. 2014 Nov;15(12):1342-50. doi: 10.1016/S1470-2045(14)70387-0. Epub 2014 Oct 1. PMID 25282284
- [Background] Kim Y, Kim YK, Lee BE, Lee SJ, Ryu YJ, Lee JH, Chang JH. Ultra-Low-Dose CT of the Thorax Using Iterative Reconstruction: Evaluation of Image Quality and Radiation Dose Reduction. AJR Am J Roentgenol. 2015 Jun;204(6):1197-202. doi: 10.2214/AJR.14.13629. PMID 26001228
- [Background] Kubo T, Ohno Y, Kauczor HU, Hatabu H. Radiation dose reduction in chest CT--review of available options. Eur J Radiol. 2014 Oct;83(10):1953-61. doi: 10.1016/j.ejrad.2014.06.033. Epub 2014 Jul 9. PMID 25066756
- [Background] Kubo T, Ohno Y, Seo JB, Yamashiro T, Kalender WA, Lee CH, Lynch DA, Kauczor HU, Hatabu H. Securing safe and informative thoracic CT examinations-Progress of radiation dose reduction techniques. Eur J Radiol. 2017 Jan;86:313-319. doi: 10.1016/j.ejrad.2016.10.012. Epub 2016 Oct 13. PMID 27773483
- [Background] Long B, Long D, Koyfman A. Emergency Medicine Evaluation of Community-Acquired Pneumonia: History, Examination, Imaging and Laboratory Assessment, and Risk Scores. J Emerg Med. 2017 Nov;53(5):642-652. doi: 10.1016/j.jemermed.2017.05.035. Epub 2017 Sep 20. PMID 28941558
- [Background] Macri F, Greffier J, Pereira F, Rosa AC, Khasanova E, Claret PG, Larbi A, Gualdi G, Beregi JP. Value of ultra-low-dose chest CT with iterative reconstruction for selected emergency room patients with acute dyspnea. Eur J Radiol. 2016 Sep;85(9):1637-44. doi: 10.1016/j.ejrad.2016.06.024. Epub 2016 Jul 1. PMID 27501900
- [Background] Martindale JL, Wakai A, Collins SP, Levy PD, Diercks D, Hiestand BC, Fermann GJ, deSouza I, Sinert R. Diagnosing Acute Heart Failure in the Emergency Department: A Systematic Review and Meta-analysis. Acad Emerg Med. 2016 Mar;23(3):223-42. doi: 10.1111/acem.12878. Epub 2016 Feb 13. PMID 26910112
- [Background] Martini K, Barth BK, Nguyen-Kim TD, Baumueller S, Alkadhi H, Frauenfelder T. Evaluation of pulmonary nodules and infection on chest CT with radiation dose equivalent to chest radiography: Prospective intra-individual comparison study to standard dose CT. Eur J Radiol. 2016 Feb;85(2):360-5. doi: 10.1016/j.ejrad.2015.11.036. Epub 2015 Dec 3. PMID 26781141
- [Background] Messerli M, Giannopoulos AA, Leschka S, Warschkow R, Wildermuth S, Hechelhammer L, Bauer RW. Diagnostic accuracy of chest X-ray dose-equivalent CT for assessing calcified atherosclerotic burden of the thoracic aorta. Br J Radiol. 2017 Dec;90(1080):20170469. doi: 10.1259/bjr.20170469. Epub 2017 Oct 3. PMID 28972810
- [Background] Messerli M, Hechelhammer L, Leschka S, Warschkow R, Wildermuth S, Bauer RW. Coronary risk assessment at X-ray dose equivalent ungated chest CT: Results of a multi-reader study. Clin Imaging. 2018 May-Jun;49:73-79. doi: 10.1016/j.clinimag.2017.10.014. Epub 2017 Oct 25. PMID 29149718
- [Background] Messerli M, Ottilinger T, Warschkow R, Leschka S, Alkadhi H, Wildermuth S, Bauer RW. Emphysema quantification and lung volumetry in chest X-ray equivalent ultralow dose CT - Intra-individual comparison with standard dose CT. Eur J Radiol. 2017 Jun;91:1-9. doi: 10.1016/j.ejrad.2017.03.003. Epub 2017 Mar 14. PMID 28629554
- [Background] Moore CL, Daniels B, Ghita M, Gunabushanam G, Luty S, Molinaro AM, Singh D, Gross CP. Accuracy of reduced-dose computed tomography for ureteral stones in emergency department patients. Ann Emerg Med. 2015 Feb;65(2):189-98.e2. doi: 10.1016/j.annemergmed.2014.09.008. Epub 2014 Nov 4. PMID 25441242
- [Background] Moser JB, Sheard SL, Edyvean S, Vlahos I. Radiation dose-reduction strategies in thoracic CT. Clin Radiol. 2017 May;72(5):407-420. doi: 10.1016/j.crad.2016.11.021. Epub 2017 Jan 27. PMID 28139204
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] O'Hora L, Foley SJ. Iterative reconstruction and automatic tube voltage selection reduce clinical CT radiation doses and image noise. Radiography (Lond). 2018 Feb;24(1):28-32. doi: 10.1016/j.radi.2017.08.010. Epub 2017 Sep 19. PMID 29306371
- [Background] Rob S, Bryant T, Wilson I, Somani BK. Ultra-low-dose, low-dose, and standard-dose CT of the kidney, ureters, and bladder: is there a difference? Results from a systematic review of the literature. Clin Radiol. 2017 Jan;72(1):11-15. doi: 10.1016/j.crad.2016.10.005. Epub 2016 Oct 31. PMID 27810168
- [Background] Ruchalski KL, Brown K. Lung Cancer Screening Update. J Thorac Imaging. 2016 Jul;31(4):190-200. doi: 10.1097/RTI.0000000000000221. PMID 27306387
- [Background] Suntharalingam S, Allmendinger T, Blex S, Al-Bayati M, Nassenstein K, Schweiger B, Forsting M, Wetter A. Spectral Beam Shaping in Unenhanced Chest CT Examinations: A Phantom Study on Dose Reduction and Image Quality. Acad Radiol. 2018 Feb;25(2):153-158. doi: 10.1016/j.acra.2017.08.011. Epub 2017 Oct 18. PMID 29055683
- [Background] Vardhanabhuti V, Pang CL, Tenant S, Taylor J, Hyde C, Roobottom C. Prospective intra-individual comparison of standard dose versus reduced-dose thoracic CT using hybrid and pure iterative reconstruction in a follow-up cohort of pulmonary nodules-Effect of detectability of pulmonary nodules with lowering dose based on nodule size, type and body mass index. Eur J Radiol. 2017 Jun;91:130-141. doi: 10.1016/j.ejrad.2017.04.006. Epub 2017 Apr 15. PMID 28629559
- [Background] Walter JE, Heuvelmans MA, de Jong PA, Vliegenthart R, van Ooijen PMA, Peters RB, Ten Haaf K, Yousaf-Khan U, van der Aalst CM, de Bock GH, Mali W, Groen HJM, de Koning HJ, Oudkerk M. Occurrence and lung cancer probability of new solid nodules at incidence screening with low-dose CT: analysis of data from the randomised, controlled NELSON trial. Lancet Oncol. 2016 Jul;17(7):907-916. doi: 10.1016/S1470-2045(16)30069-9. Epub 2016 Jun 6. PMID 27283862
- [Background] Yousaf-Khan U, van der Aalst C, de Jong PA, Heuvelmans M, Scholten E, Lammers JW, van Ooijen P, Nackaerts K, Weenink C, Groen H, Vliegenthart R, Ten Haaf K, Oudkerk M, de Koning H. Final screening round of the NELSON lung cancer screening trial: the effect of a 2.5-year screening interval. Thorax. 2017 Jan;72(1):48-56. doi: 10.1136/thoraxjnl-2016-208655. Epub 2016 Jun 30. PMID 27364640
- [Background] Yousaf-Khan U, van der Aalst C, de Jong PA, Heuvelmans M, Scholten E, Walter J, Nackaerts K, Groen H, Vliegenthart R, Ten Haaf K, Oudkerk M, de Koning H. Risk stratification based on screening history: the NELSON lung cancer screening study. Thorax. 2017 Sep;72(9):819-824. doi: 10.1136/thoraxjnl-2016-209892. Epub 2017 Mar 30. PMID 28360223
- [Background] Zinsser D, Marcus R, Othman AE, Bamberg F, Nikolaou K, Flohr T, Notohamiprodjo M. Dose Reduction and Dose Management in Computed Tomography - State of the Art. Rofo. 2018 Jun;190(6):531-541. doi: 10.1055/s-0044-101261. Epub 2018 Mar 13. PMID 29534253
- [Derived] Wassipaul C, Janata-Schwatczek K, Domanovits H, Tamandl D, Prosch H, Scharitzer M, Polanec S, Schernthaner RE, Mang T, Asenbaum U, Apfaltrer P, Cacioppo F, Schuetz N, Weber M, Homolka P, Birkfellner W, Herold C, Ringl H. Ultra-low-dose CT vs. chest X-ray in non-traumatic emergency department patients - a prospective randomised crossover cohort trial. EClinicalMedicine. 2023 Oct 17;65:102267. doi: 10.1016/j.eclinm.2023.102267. eCollection 2023 Nov. PMID 37876998
- See also: Austrian Federal Ministry of Labour, Social Affairs, Health and Consumer Protection 2018a. Radiation Application in Medicine | Health Portal [Online]. [Accessed: 22 November 2018]. — https://www.gesundheit.gv.at/leben/umwelt/radiokativitaet/medizin
- See also: Austrian Federal Ministry of Labour, Social Affairs, Health and Consumer Protection 2018b. Radiation Exposure in Austria | Health Portal [Online]. [Accessed: 22 November — https://www.gesundheit.gv.at/leben/umwelt/radiokativitaet/strahlenbelastung
- See also: German Federal Office for Radiation Protection. Diagnostic Reference Levels. June 2016 — https://www.bfs.de/SharedDocs/Downloads/BfS/DE/fachinfo/ion/drw-roentgen.pdf?__blob=publicationFile&v=9
- See also: Gesundheit Österreich GmbH (Health Austria GmbH). Update on diagnostic reference values for Austria 2017 — https://jasmin.goeg.at/384/1/Aktualisierung%20der%20diagnostischen%20Referenzwerte_0-Fehler.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03922516/Prot_SAP_002.pdf
  • Informed Consent Form (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/16/NCT03922516/ICF_003.pdf